CLINICAL TRIAL: NCT07097376
Title: Evaluating the Efficacy of a Vocational Counseling Intervention to Improve Occupational Functioning and Employment Quality Among Veterans With Mental Health and Substance Use Disorders
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: North Texas Veterans Healthcare System (U.S. Federal Agency); VA Hines Health Care (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RRD4-001-24W
Record Dates: First submitted 2025-07-16; First posted 2025-07-31 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Unemployment
Keywords: rehabilitation, vocational

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to either a treatment as usual condition or to receive treatment as usual along with the additional intervention of Purposeful Pathways.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Purposeful Pathways (Experimental): Participants in this arm will receive treatment as usual, which is the transitional work intervention, as well as the Purposeful Pathways intervention
  Interventions: Behavioral: Purposeful Pathways; Other: Transitional Work
- Treatment as usual (Active Comparator): Participants in this arm will receive treatment as usual, which is the transitional work intervention.
  Interventions: Other: Transitional Work

INTERVENTIONS:
Behavioral: Purposeful Pathways — Purposeful Pathways is a manualized intervention to assist Veterans in aspiring and pursuing meaningful employment. Purposeful Pathways is an individual counseling protocol delivered weekly for up to 12 sessions (50 minutes per session) focused on career exploration, goal clarity, job-searching, and self-regulation.
  Arms: Purposeful Pathways
Other: Transitional Work — Provides individuals with immediate access to a non-competitive, paid job contracted by the VA. Positions are typically housed within a VA hospital (e.g., housekeeping, grounds, kitchens, and construction), but are sometimes located in the community. TW is time-limited. TW is staffed by vocational rehabilitation specialists (VRS).
  Other Names: CWT

SUMMARY:
Veterans living with mental health and substance use conditions are at risk of unemployment, which leads to significant health-related consequences. Though the Veterans Health Administration offers numerous vocational rehabilitation programs to address unemployment, they are not uniformly effective for everyone who participates. This project will test a new model for addressing Veteran unemployment. This new model adds career development services (a vocational counseling program called Purposeful Pathways) to a standard model of vocational rehabilitation (a program called Transitional Work [TW]). The investigators will test if adding Purposeful Pathways to TW leads to more Veterans working in quality jobs as well as better quality of life, reduced mental health symptoms, and reduced substance use. This project fills a critical need in advancing research and practice aimed at reducing Veteran unemployment; thereby preventing consequences to Veteran's economic, social, and health related functioning and well-being.

The investigators will conduct a phase II, multi-site, RCT comparing Purposeful Pathways + TW (n=127) to TW alone (n=127) among Veterans participating in TW at VA Bedford, VA Hines, and VA North Texas. Aim 1: Evaluate the efficacy of Purposeful Pathways for improving occupational functioning (primary outcome). Hypothesis: Purposeful Pathways + TW, compared to TW only, will improve occupational functioning. Aim 2: Evaluate the efficacy of Purposeful Pathways for improving quality of life, and reducing mental health symptoms and substance use (secondary outcomes). Hypothesis: Purposeful Pathways + TW, compared to TW only, will improve quality of life, and reduce mental health symptoms and substance use. Aim 3 (Exploratory): Explore whether occupational functioning (competitive employment attainment) in the Purposeful Pathways + TW group is mediated by vocational identity, work hope, self-regulation, and/or employment motivation, key factors central to the Purposeful Pathways intervention.

DETAILED DESCRIPTION:
The investigators will conduct a multi-site efficacy RCT comparing Purposeful Pathways + transitional work (TW) (n=127) to TW alone (n=127) with sites at VA Bedford (Bedford, MA), VA Hines (Chicago, IL), and VA North Texas (Dallas, TX). The proposed project will allow us to evaluate the efficacy of Purposeful Pathways as an augmentation to TW for improving the primary outcome of occupational functioning, as well as downstream improvements in secondary outcomes of quality of life, mental health, and substance use. The investigators will also explore whether occupational functioning outcomes in the Purposeful Pathways + TW group are mediated by the factors proposed by the underlying theoretical model for Purposeful Pathways.

Aim 1: Evaluate the efficacy of Purposeful Pathways for improving occupational functioning (primary outcomes) Hypothesis 1a-e: Purposeful Pathways + TW, compared to TW only, will improve occupational functioning at a 12-month follow-up as evidenced by (1a) rates of competitive employment, (1b) hours worked, (1c) income earned, (1d) career adaptabilities (Career Adapt-Abilities Scale), and (1e) meaningful employment (Work as Meaning Inventory-Positive Meaning Subscale).

Aim 2: Evaluate the efficacy of Purposeful Pathways for improving quality of life, and reducing mental health symptoms and substance use (secondary outcomes) Hypothesis 2a-c: Purposeful Pathways + TW, compared to TW only, will improve (2a) quality of life (Quality of Life Enjoyment and Satisfaction Questionnaire-Short Form), and reduce (2b) mental health symptoms (Patient Health Questionnaire) and (2c) substance use (Tobacco, Alcohol, Prescription medications, and other Substance tool) at a 12-month follow-up

Aim 3 (Exploratory): Explore whether occupational functioning (competitive employment attainment) in the Purposeful Pathways + TW group is mediated by vocational identity, work hope, self-regulation, and/or employment motivation, key factors central to the Purposeful Pathways intervention.

The study intervention is a behavioral intervention. Purposeful Pathways is a manualized, vocational counseling intervention based on a Veteran-centered, recovery-oriented approach. The overarching target of the intervention is to increase motivation to pursue meaningful employment goals by enhancing vocational identity/positive vocational self-appraisals, increasing work hope (goals, pathways, and self-efficacy), and promoting employment-related self-regulation skills. The table below provides an overview of the specific treatment elements associated with each of the four core components: 1) career/identity exploration, 2) goal setting/planning, 3) job-search skill building, and 4) self-regulation skill building. The Purposeful Pathways intervention will be provided over 12 weeks by a master's level clinician affiliated with their respective (Bedford, Hines, of North Texas) vocational rehabilitation program. Sessions will be provided in person or through the VHA telehealth services platform (VVC).

All participants will complete the following surveys/questionnaires.

Demographics. The investigators will gather basic demographic information including age, gender, race, level of education, service-connected percentage, service connected condition, receipt of disability pensions, housing stability, and history of substance abuse and mental health diagnoses.

Competitive employment. The investigators will ask whether a Veteran has been competitively employed at any point over the previous month. In line with other RCT research, the investigators define competitive employment as "a non-sheltered job earning salary, wages, or commission, excluding military drill and transient cash-based jobs, such as yard work, babysitting, and manual day labor." (p. 318). For those employed, the investigators will also ask for job title, industry, and company names.

Weeks/hours worked. Among those who have worked in a competitive job, we will ask about the number of days/weeks worked over the past month, as well as the number of hours worked.

Income earned. Among those who have worked in a competitive job, the investigators will ask for the participants' hourly wage.

Career-related adaptability skills. The Career Adapt-Abilities Scale (CAAS) will be utilized to measure one's level of career adaptability, a commonly used measure of ability and skill for navigating long-term career advancement. This is a 24-item measure that is grouped into four different subscales that capture total adaptability along with four dimensions: concern, control, curiosity, and confidence. Respondents are asked to rate how strongly they have developed each of these strengths using a 5-point Likert type scale. Responses range from 5 ("Strongest") to 1 ("Not strong").

Meaningful employment. The Positive Meaning Scale of the Work as Meaning Inventory (WAMI) will be used to measure the degree to which someone perceives their work as meaningful. The Positive Meaning scale consists of 4 items answered on a 7-point scale ranging from 1 (strongly disagree) to 7 (strongly agree). Higher scores represent higher levels of meaningful work. This scale has been used extensively in the vocational literature and has demonstrated consistent reliability and validity, including with Veterans with co-occurring conditions.

Job-Searching Behavior. The Job-Search Intensity Scale (JSIS) will be utilized to assess the level of time one spent on various job-search activities. This nine-item measure asks respondents about the following job-search activities: preparing/revising resume, reading classified/help. wanted advertisements, looking for jobs on the Internet, talking with friends/relatives about job leads, speaking with previous employers or business acquaintances about job leads, contacting employment agencies, making inquiries to prospective employers, sending out application letters, and preparing and going on job interviews. Responses to each activity are measured on a 5-point, Likert-type scale to assess the amount of time spent on each activity. Possible scores for each item range from 1 ("No time at all") to 5 ("Very much time").

Quality of life. The Quality of Life Enjoyment and Satisfaction Questionnaire - Short Form (Q-LES-Q - SF) will be used as a measure of general psychiatric functioning. The Q-LES-Q - SF is a 16 item self-report measure of perceived functioning and is one of the most widely used outcomes measures in psychiatric research.

Mental health: The Patient Health Questionnaire-9 (PHQ-9) is a 9-item measure of common mental health symptoms associated with depression. It is a widely used and available inventory in VHA with good validity and reliability.

Substance use. Substance use outcomes include frequency, quantity, and severity of substance use, and will be measured with the Tobacco, Alcohol, Prescription medications, and other Substance (TAPS) tool, which is used within the National Institute on Drug Abuse (NIDA) clinical trials network.

Vocational identity. The Vocational Identity Scale (VIS) will measure the extent to which an individual possesses a clear and stable understanding of his or her goals, interests, and talents as related to vocational decisions. The VIS consists of 18 true or false items that asks respondents to identify whether the statement is mostly "True" or mostly "False." Higher scores indicate more crystallized vocational identity. The VIS is extensively used in vocational psychology literature and has undergone psychometric analysis demonstrating validity and reliability, and has been used in studies with Veterans and those with psychiatric disorders.

Work hope. The Work Beliefs Scale (WBS) will be utilized to measure work hope. This is a 24-item measure on a seven-point scale ranging from "Strongly disagree" to "strongly agree." Respondents are asked to rate their level of agreement on various items empirically related to work hope (having a goal, having a plan to reach goal, and having self-efficacy to pursue one's goal). Validity and reliability among individuals with significant psychosocial barriers have been established.

Self-regulation. The Short Self-Regulation Questionnaire (SSRQ) will be used to measure self-regulation skills. This 31-item self-report measures asks respondents to respond to items on a 5 point Likert type scale ranging from strongly disagree to strongly agree. The measure demonstrated construct validity and demonstrated high internal consistency among Veterans with co-occurring conditions.

Employment motivation. The Importance of Obtaining Preferred Position (IOPP) will be used to measure motivational attitudes to attain preferred employment. This is a 5-item measure on a five-point scale ranging from "Not important" to "Very Important." This scale has been validated and has been used widely in vocational literatures as an measure of motivational commitment to employment among individuals who are unemployed.

Client satisfaction. The Client Satisfaction Questionnaire-8 (CSQ-8) will be used to measure satisfaction, perceived quality, and effectiveness of treatment. This self-report questionnaire consists of eight items, scored 1 to 4, with higher scores indicating higher satisfaction with treatment. The CSQ-8 has been used in mental health and other health centers and has acceptable internal consistency.

Exit interviews. The investigators will randomly ask 30 Veterans participating in the intervention arm to complete a brief qualitative exit interview (15-minutes) at 12-week treatment end. These semi-structured, open-ended interviews will take place via phone, VVC, or in-person depending on Veteran's preference. Questions will assess barriers and facilitators of treatment engagement (e.g., Describe how the timing of the intervention fit into your day/week and overall recovery. Would you recommend the intervention earlier or later in your recovery? Would you recommend the intervention as in-person or virtual? Were there issues being able to attend your appointments? Did you received any feedback from your TW counselor or workplace supervisor about attending appointments?). Interviews will be recorded via VA-approved recording technologies and will be transcribed by a VA-approved transcription service.

ELIGIBILITY:
Inclusion Criteria:

* enrolled in VHA TW at one of the three VA recruitment sites
* be unemployed
* report interest/intention to return to paid work within the upcoming three years
* presence of a psychiatric disorder as indicated by documented ICD-10 diagnosis (mental health disorder and/or substance use disorder) addressed in an encounter at VHA within the 24 months preceding study enrollment
* ages 18 and over
* willing to participate in weekly vocational counseling sessions

Exclusion Criteria:

* report a plan to remain unemployed during the upcoming 12 months
* report plans to retire within the next 12 months
* be currently retired
* be a full-time student
* enrolled in Supported Employment
* experiencing significantly elevated mental health symptoms as indicated by a score greater than 26 on the Symptom Checklist-6 (SCL-648)
* have a guardian or conservator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 254 (Estimated)
Dates: Start 2026-05-01 (Estimated); Primary Completion 2030-10-01 (Estimated); Study Completion 2031-03-31 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Competitive Employment | through study completion, an average of 15 months
  Number of participants who were competitively employed at any point over the previous month. We define competitive employment as a non-sheltered job that earns salary, wages, or commission, excluding military drill and transient cash-based jobs, such as yard work, babysitting, and manual day labor.
Number of days worked | through study completion, an average of 15 months
  The number of days worked in competitive employment over the past month
Total hours worked | through study completion, an average of 15 months
  The number of hours worked in competitive employment during previous month
Income earned | through study completion, an average of 15 months
  Total wages from competitive employment earned over the past month
Career Adapt-Ability Scale | through study completion, an average of 15 months
  One's functional abilities/strengths to successfully manage career-related tasks. Possible scores range from 24 - 120, with greater scores indicating greater career adaptability functioning.
Positive Meaning Scale of the Work as Meaning Inventory | through study completion, an average of 15 months
  Degree to which someone perceives their work as meaningful. Scores range from 4 - 28, with higher scores representing greater levels of meaningful work.

SECONDARY OUTCOMES:
Quality of Life Enjoyment and Satisfaction Questionnaire-Short Form | through study completion, an average of 15 months
  A self-report measure of perceived functioning. Scores range from 14 - 70 with higher scores indicating greater perceived functioning
Patient Health Questionnaire-9 | through study completion, an average of 15 months
  Mental health symptom inventory. Responses range from 0 - 27, with greater scores indicating more severe mental health symptoms.
Alcohol misuse | through study completion, an average of 15 months
  The Tobacco, Alcohol, Prescription medications, and other Substance (TAPS) Tool Part 2 will assess alcohol misuse in the past three months. This scale consists of four Yes or No items (Yes = 1 and No = 0). Scores range from 0 - 4, with greater scores indicating greater alcohol misuse.
Marijuana misuse | through study completion, an average of 15 months
  The Tobacco, Alcohol, Prescription medications, and other Substance (TAPS) Tool Part 2 will assess marijuana misuse in the past three months. This scale consists of three Yes or No items (Yes = 1 and No = 0). Scores range from 0 - 3, with greater scores indicating greater marijuana misuse.
Cocaine, crack, or methamphetamine misuse | through study completion, an average of 15 months
  The Tobacco, Alcohol, Prescription medications, and other Substance (TAPS) Tool Part 2 will assess cocaine, crack, or methamphetamine misuse in the past three months. This scale consists of three Yes or No items (Yes = 1 and No = 0). Scores range from 0 - 3, with greater scores indicating greater cocaine, crack, or methamphetamine misuse.
Heroin misuse | through study completion, an average of 15 months
  The Tobacco, Alcohol, Prescription medications, and other Substance (TAPS) Tool Part 2 will assess heroin misuse in the past three months. This scale consists of three Yes or No items (Yes = 1 and No = 0). Scores range from 0 - 3, with greater scores indicating greater heroin misuse.
Prescription opiate misuse | through study completion, an average of 15 months
  The Tobacco, Alcohol, Prescription medications, and other Substance (TAPS) Tool Part 2 will assess prescription opiate misuse in the past three months. This scale consists of three Yes or No items (Yes = 1 and No = 0). Scores range from 0 - 3, with greater scores indicating greater prescription opiate misuse.
Medication for anxiety or sleep misuse | through study completion, an average of 15 months
  The Tobacco, Alcohol, Prescription medications, and other Substance (TAPS) Tool Part 2 will assess medication for anxiety or sleep misuse in the past three months. This scale consists of three Yes or No items (Yes = 1 and No = 0). Scores range from 0 - 3, with greater scores indicating greater medication for anxiety or sleep misuse.
Medication for ADHD misuse | through study completion, an average of 15 months
  The Tobacco, Alcohol, Prescription medications, and other Substance (TAPS) Tool Part 2 will assess medication for ADHD misuse in the past three months. This scale consists of three Yes or No items (Yes = 1 and No = 0). Scores range from 0 - 3, with greater scores indicating greater medication for ADHD misuse.
Other illegal or recreational drug use | through study completion, an average of 15 months
  The Tobacco, Alcohol, Prescription medications, and other Substance (TAPS) Tool Part 2 will assess any other illegal or recreational drug (for example, ecstasy/molly, GHB, poppers, LSD, mushrooms, special K, bath salts, synthetic marijuana ('spice'),whip-its, etc.) in the past three months. This is a single item Yes or No question (Yes = 1 and No = 0). Scores range from 0 - 1, with greater scores indicating use of other illegal or recreational drugs.

OTHER OUTCOMES:
Vocational identity scale | through study completion, an average of 15 months
  Self-report measure of the extent to which an individual possesses a clear and stable understanding of his or her goals, interests, and talents as related to vocational decisions (i.e., vocational identity). The scale consists of 18 true or false items that asks respondents to identify whether the statement is mostly "True" or mostly "False." Higher scores indicate better vocational identity.
Work Beliefs Scale | through study completion, an average of 15 months
  Self-report measure of work-related hope. Scores range from 24 - 168 with greater scores indicating greater work hope.
Short Self-Regulation Questionnaire | through study completion, an average of 15 months
  Self-report measure of self-regulation skills. Scores range from 31 - 155, with higher scores indicating greater self-regulation skills.
Importance of Obtaining Preferred Position Scale | through study completion, an average of 15 months
  Self-report motivational attitudes toward attaining employment. Scores range from 5 - 25 and higher scores indicate greater motivation to obtain employment.
Job Search Intensity Scale | through study completion, an average of 15 months
  This self-report measure assesses the level of time one spent on various job-search activities. Scores range from 9 - 45 with higher scores indicating greater engagement in job-search behaviors.
Client Satisfaction Questionnaire-8 (CSQ-8) | end of treatment phase (week 12)
  Measure of client satisfaction with treatment received. Scores range from 8 - 32 with high scores indicating greater satisfaction with treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Brian J Stevenson, PhD, Principal Investigator — VA Bedford HealthCare System, Bedford, MA
Locations (3):
- United States (3):
  - Edward Hines Jr. VA Hospital, Hines, IL, Hines, Illinois
  - VA Bedford HealthCare System, Bedford, MA, Bedford, Massachusetts
  - VA North Texas Health Care System Dallas VA Medical Center, Dallas, TX, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No